CLINICAL TRIAL: NCT00828139
Title: A Randomized Phase II Trial of Weekly Topotecan With and Without AVE0005 (Aflibercept; NSC-724770) in Patients With Platinum Treated Extensive Stage Small Cell Lung Cancer (E-SCLC)
Brief Title: S0802 - Topotecan With or Without Aflibercept in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01182; NCI-2009-01182 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0802; CDR0000632614; S0802 (Other: Southwest Oncology Group); S0802 (Other: CTEP)
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — aflibercept; Topotecan; trioctyl phosphine oxide

ARMS (2):
- Arm I (ziv-aflibercept, topotecan hydrochloride) (Experimental): Patients receive ziv-aflibercept IV over 1 hour on day 1 and topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responsive or stable disease after 4 courses may then receive ziv-aflibercept IV on day 1 and topotecan hydrochloride IV on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept; Drug: topotecan hydrochloride
- Arm II (topotecan hydrochloride) (Active Comparator): Patients receive topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responsive or stable disease after 4 courses may then receive topotecan hydrochloride IV on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: topotecan hydrochloride

INTERVENTIONS:
Biological: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap
  Arms: Arm I (ziv-aflibercept, topotecan hydrochloride)
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO

SUMMARY:
This randomized phase II trial is studying topotecan to see how well it works when given with or without aflibercept in treating patients with extensive-stage small cell lung cancer. Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Combinations of biological substances in aflibercept may be able to carry tumor-killing substances directly to small cell lung cancer cells. Aflibercept may also stop the growth of small cell lung cancer by blocking blood flow to the tumor. It is not yet known whether topotecan is more effective with or without aflibercept in treating patients with small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the efficacy of topotecan hydrochloride with vs without aflibercept (ziv-aflibercept), in terms of progression-free survival at 3 months, in patients with extensive stage small cell lung cancer previously treated with platinum-based therapy.

SECONDARY OBEJCTIVES:

I. Assess the response rate (confirmed and unconfirmed, complete and partial responses) in a subset of patients with measurable disease.

II. Assess the overall survival of these patients. III. Evaluate the frequency and severity of toxicities of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to response to prior platinum-based therapy (platinum-sensitive disease vs platinum-refractory disease). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive ziv-aflibercept IV over 1 hour on day 1 and topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responsive or stable disease after 4 courses may then receive ziv-aflibercept IV on day 1 and topotecan hydrochloride IV on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responsive or stable disease after 4 courses may then receive topotecan hydrochloride IV on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive stage small cell lung cancer

  * Progressive or recurrent disease following one (and only one) standard first-line platinum-containing regimen (cisplatin or carboplatin)
* Measurable or non-measurable disease per RECIST criteria

  * Disease must be outside a previously irradiated field OR a new lesion must be inside the irradiated field
  * Disease must be outside a previously resected area OR a new lesion must be present
* No known brain metastasis unless the metastasis has been treated and is stable for ≥ 3 months prior to study entry
* No leptomeningeal involvement or brain stem metastasis
* Zubrod performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal OR creatinine clearance ≥ 60 mL/min
* Urine protein: creatinine ratio < 1 OR urine protein < 500 mg by 24-hour urine collection
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Willing to provide smoking history
* No evidence of active infection
* No active bleeding
* No significant history of bleeding diathesis, including hemoptysis (½ teaspoon of hemoptysis within the past 3 months), or underlying coagulopathy
* No history of recent arterial embolic events, including any of the following:

  * Myocardial infarction
  * Cerebrovascular accident
  * Transient ischemic attack
  * Worsening of pre-existing angina within the past 6 months
* No uncontrolled hypertension (systolic BP > 150 mm Hg or diastolic BP > 100 mm Hg)

  * History of hypertension allowed provided it is controlled on anti-hypertensive medications
* No history of congestive heart failure
* No history of encephalitis or encephalopathy of any cause
* No diverticulitis, gastrointestinal bleeding, or peptic ulcer within the past 3 months
* No known AIDS or HIV-1 associated complex
* No known history of immune or immunodeficiency disorders
* No unstable or pre-existing major medical conditions except for cancer-related abnormalities
* No other prior malignancy except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer currently in complete remission
  * Any other cancer from which the patient been disease-free for 5 years
* Concurrent chronic therapeutic doses of low molecular weight heparin allowed
* At least 21 days since prior and no concurrent radiotherapy and recovered
* At least 28 days since prior and no concurrent surgery (e.g., thoracic or other major surgeries) and recovered
* No prior bevacizumab or other anti-angiogenic therapies including, but not limited to, small molecule tyrosine kinase inhibitors
* No concurrent enzyme-inducing anticonvulsant drugs

  * Non-enzyme-inducing anticonvulsant drugs (e.g., Keppra) allowed
* Concurrent chronic oral anticoagulation therapy allowed provided INR is maintained in the therapeutic range (INR 2-3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Allen, Principal Investigator — SWOG Cancer Research Network
Locations (257):
- United States (257):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Providence Hospital, Mobile, Alabama
  - Arizona Cancer Center at UMC Orange Grove, Tucson, Arizona
  - Arizona Cancer Center at University Medical Center North, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group-Rogers, Rogers, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope Medical Center, Duarte, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institute CCOP, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - University of California at Davis Cancer Center, Sacramento, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Hays Medical Center, Hays, Kansas
  - Promise Regional Medical Center-Hutchinson, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas City Cancer Center-West, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Ozark Health Ventures LLC dba Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Arnot Ogden Medical Center, Elmira, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University Medical Center, New York, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Carolinas Medical Center - Northeast, Concord, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - AnMed Health Hospital, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee - Memphis, Memphis, Tennessee
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Saint Luke's Episcopal Hospital, Houston, Texas
  - Veterans Administration Medical Center, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Southwest Oncology Group, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Lara PN Jr, Moon J, Redman MW, Semrad TJ, Kelly K, Allen JW, Gitlitz BJ, Mack PC, Gandara DR. Relevance of platinum-sensitivity status in relapsed/refractory extensive-stage small-cell lung cancer in the modern era: a patient-level analysis of southwest oncology group trials. J Thorac Oncol. 2015 Jan;10(1):110-5. doi: 10.1097/JTO.0000000000000385. PMID 25490004
- [Derived] Allen JW, Moon J, Redman M, Gadgeel SM, Kelly K, Mack PC, Saba HM, Mohamed MK, Jahanzeb M, Gandara DR. Southwest Oncology Group S0802: a randomized, phase II trial of weekly topotecan with and without ziv-aflibercept in patients with platinum-treated small-cell lung cancer. J Clin Oncol. 2014 Aug 10;32(23):2463-70. doi: 10.1200/JCO.2013.51.4109. Epub 2014 Jul 7. PMID 25002722

RESULTS

PARTICIPANT FLOW:
Groups:
- Platinum-Sensitive Treated With Topotecan and Ziv-aflibercept: Patients with platinum sensitive (complete response or partial response and > 90 day treatment-free interval for extensive stage or ≥ 180 days for limited stage) were treated with Topotecan and ziv-aflibercept.
- Platinum Sensitivity Treated With Topotecan Alone: Patients with platinum sensitivity treated with topotecan alone
- Platinum Refractory Treated With Topotecan + Ziv-aflibercept: Patients with platinum refractory (no response and/or treatment-free interval ≤ 90 days for extensive stage and < 180 days for limited stage) treated topotecan and ziv-aflibercept.
- Platinum Refractory Treated With Topotecan Aloine: Patients with platinum refractory treated topotecan alone.
Period: Overall Study
Arm/Group | Platinum-Sensitive Treated With Topotecan and Ziv-aflibercept | Platinum Sensitivity Treated With Topotecan Alone | Platinum Refractory Treated With Topotecan + Ziv-aflibercept | Platinum Refractory Treated With Topotecan Aloine
Started | 42 | 41 | 55 | 51
Completed | 1 | 0 | 0 | 0
Not Completed | 41 | 41 | 55 | 51
Not completed — Adverse Event | 8 | 1 | 10 | 5
Not completed — Death | 2 | 1 | 0 | 2
Not completed — Refusal unrelated to toxicity | 3 | 4 | 5 | 3
Not completed — Disease Progression | 24 | 33 | 35 | 39
Not completed — Other | 4 | 2 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platinum-Sensitive Treated With Topotecan and Ziv-aflibercept | Platinum Sensitivity Treated With Topotecan Alone | Platinum Refractory Treated With Topotecan + Ziv-aflibercept | Platinum Refractory Treated With Topotecan Aloine | Total
Number analyzed (Participants) | 42 | 41 | 55 | 51 | 189
Age, Continuous [Median (Full Range); unit: years] | 63.4 [43.1 to 81.8] | 60.1 [33.2 to 85.1] | 60.9 [40.1 to 82.6] | 63.6 [45.1 to 85.1] | 62.5 [33.2 to 85.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 29 | 17 | 99
  Male | 17 | 13 | 26 | 34 | 90
Race/Ethnicity, Customized [Number; unit: participants]
  White | 36 | 40 | 49 | 43 | 168
  Black | 4 | 1 | 3 | 4 | 12
  Pacific Islander | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1
  Native American | 0 | 0 | 2 | 1 | 3
  Unknown/Other | 1 | 0 | 1 | 2 | 4
Metastatic Disease Sites [Number; unit: participants]
  Single lesion, single organ | 4 | 9 | 4 | 4 | 21
  Multiple lesions, single organ | 11 | 9 | 9 | 11 | 40
  Multiple lesions, multiple organs | 25 | 22 | 41 | 34 | 122
  None | 2 | 1 | 1 | 2 | 6
Stage [Number; unit: participants] — In limited stage small cell lung cancer, the cancer resides in one lung or in the nearby tissue.
  In the extensive stage, cancer has spread to tissue outside of the originally affected lung.
  participants
    Extensive | 27 | 23 | 39 | 42 | 131
    Limited | 15 | 18 | 16 | 9 | 58
Performance Status [Number; unit: participants] — 0 ----- Fully active, able to carry on all pre-disease performance without restriction.
  1 ----- Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  The higher grade, the worse outcome.
  participants
    0 | 14 | 17 | 12 | 19 | 62
    1 | 28 | 24 | 43 | 32 | 127

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: From the date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause.
  Progression is defined as 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: Disease assessments were performed every 6 weeks, up to 2 years.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Platinum-Sensitive Treated With Topotecan and Ziv-aflibercept | Platinum Sensitivity Treated With Topotecan Alone | Platinum Refractory Treated With Topotecan + Ziv-aflibercept | Platinum Refractory Treated With Topotecan Aloine
Number analyzed (Participants) | 42 | 41 | 55 | 51
Months | 1.8 [1.5 to 2.2] | 1.3 [1.2 to 1.4] | 1.4 [1.3 to 1.7] | 1.4 [1.3 to 1.4]
Statistical Analysis 1: Comparison: Platinum-Sensitive Treated With Topotecan and Ziv-aflibercept; 3-month PFS was estimated using the method of Kaplan-Meier. The 3-month PFS estimated value corresponds to the probability of PFS at month 3; Test type: Superiority or Other; 3-month PFS = 0.24, 90% CI 2-sided [0.14 to 0.37] — The estimated value corresponds to the probability of PFS at month 3
Statistical Analysis 2: Comparison: Platinum Sensitivity Treated With Topotecan Alone; 3-month PFS was estimated using the method of Kaplan-Meier; Test type: Superiority or Other; 3-month PFS = 0.15, 90% CI 2-sided [0.07 to 0.27] — The estimated value corresponds to the probability of PFS at month 3
Statistical Analysis 3: Comparison: Platinum Refractory Treated With Topotecan + Ziv-aflibercept; 3-month PFS was estimated using the method of Kaplan-Meier; Test type: Superiority or Other; 3-month PFS = 0.27, 90% CI 2-sided [0.18 to 0.39] — The estimated value corresponds to the probability of PFS at month 3
Statistical Analysis 4: Comparison: Platinum Refractory Treated With Topotecan Aloine; 3-month PFS was estimated using the method of Kaplan-Meier; Test type: Superiority or Other; 3-month PFS = 0.1, 90% CI 2-sided [0.04 to 0.2] — The estimated value corresponds to the probability of PFS at month 3
Statistical Analysis 5: Comparison: Platinum-Sensitive Treated With Topotecan and Ziv-aflibercept vs Platinum Sensitivity Treated With Topotecan Alone; Hazard Ratio was evaluated using a logrank test; Test type: Superiority or Other; Hazard Ratio (HR) = 1.32, 90% CI 2-sided [0.91 to 1.92]
Statistical Analysis 6: Comparison: Platinum Refractory Treated With Topotecan + Ziv-aflibercept vs Platinum Refractory Treated With Topotecan Aloine; Hazard Ratio was evaluated using log-rank test; Test type: Superiority or Other; Hazard Ratio (HR) = 1.51, 90% CI 2-sided [1.08 to 2.10]

2. Secondary Outcome: Overall Survival
Description: Estimated to within at least 15% (95% confidence interval).
Time Frame: Weekly, up to 2 years.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Platinum-Sensitive Treated With Topotecan and Ziv-aflibercept | Platinum Sensitivity Treated With Topotecan Alone | Platinum Refractory Treated With Topotecan + Ziv-aflibercept | Platinum Refractory Treated With Topotecan Aloine
Number analyzed (Participants) | 42 | 41 | 55 | 51
months | 6.0 [4.8 to 10.2] | 4.6 [2.9 to 5.3] | 4.6 [4.0 to 5.8] | 4.2 [2.7 to 5.0]

3. Secondary Outcome: Response Rate (Confirmed and Unconfirmed, Complete and Partial Responses)
Description: The number of confirmed and unconfirmed complete and partial responses in the subset of patients with measurable disease per RECIST 1.0. Estimated to within at least 17% (95% confidence interval).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Disease assessment for response were performed every 6 weeks, up to 2 years.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Platinum-Sensitive Treated With Topotecan and Ziv-aflibercept | Platinum Sensitivity Treated With Topotecan Alone | Platinum Refractory Treated With Topotecan + Ziv-aflibercept | Platinum Refractory Treated With Topotecan Aloine
Number analyzed (Participants) | 41 | 39 | 51 | 48
proportion of participants | 0.02 [0 to 0.11] | 0 [0 to 0.07] | 0.02 [0 to 0.09] | 0 [0 to 0.06]

4. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 3.0. Only adverse events that are possibly, probably or definitely related to study drug are reported. The events listed here are not necessary to be included in Serious Adverse Event. A serious event could be death, life-threatening, hospitalization, disability or permanent damage, congenital anomaly...Grade 3 through 5 adverse event may not meet the criterion of serious adverse event.
Time Frame: Toxicity assessment was evaluated after each cycle (21 days), up to 2 years.
Population: Eligible patients who had received the protocol treatments were included in the adverse event summaries. Ant CTCAE 3.0 event of Grade 3 (serious), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Ziv-aflibercept + Topotecan | Topotecan
Number analyzed (Participants) | 92 | 87
Participants
  AST, SGOT | 1 | 2
  Anorexia | 3 | 2
  Bilirubin (hyperbilirubinemia) | 1 | 0
  Bronchospasm, wheezing | 0 | 1
  Calcium, serum-high (hypercalcemia) | 1 | 0
  Cardiac-ischemia/infarction | 1 | 0
  Colitis, infectious (e.g., Clostridium difficile) | 1 | 0
  Confusion | 3 | 0
  Constipation | 0 | 1
  Creatinine | 0 | 1
  Dehydration | 6 | 1
  Diarrhea | 1 | 0
  Dizziness | 2 | 1
  Dyspnea (shortness of breath) | 7 | 1
  Fatigue (asthenia, lethargy, malaise) | 15 | 3
  Febrile neutropenia | 1 | 0
  GGT (gamma-glutamyl transpeptidase) | 1 | 0
  Hemoglobin | 9 | 7
  Hemolysis | 1 | 1
  Hemorrhage, GI - Upper GI NOS | 2 | 0
  Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS | 1 | 0
  Hemorrhage, pulmonary/upper respiratory - Lung | 1 | 0
  Hemorrhage, pulmonary/upper respiratory - Nose | 2 | 0
  Hypertension | 3 | 0
  INR (of prothrombin time) | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Colon | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 0 | 1
  Infection with unknown ANC - Blood | 0 | 2
  Infection with unknown ANC - Lung (pneumonia) | 1 | 0
  Left ventricular systolic dysfunction | 1 | 0
  Leukocytes (total WBC) | 17 | 22
  Leukoencephalopathy (radiolographic findings) | 1 | 0
  Lipase | 1 | 0
  Lymphopenia | 5 | 13
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1 | 0
  Muscle weakness, not d/t neuropathy - body/general | 3 | 1
  Nausea | 4 | 1
  Neutrophils/granulocytes (ANC/AGC) | 30 | 23
  Pain - Abdomen NOS | 3 | 0
  Pain - Chest wall | 1 | 0
  Pain - Head/headache | 2 | 0
  Pain - Pain NOS | 1 | 0
  Platelets | 29 | 17
  Pneumonitis/pulmonary infiltrates | 0 | 1
  Potassium, serum-high (hyperkalemia) | 0 | 1
  Potassium, serum-low (hypokalemia) | 3 | 1
  Proteinuria | 1 | 0
  Psychosis (hallucinations/delusions) | 0 | 1
  Renal failure | 0 | 2
  Seizure | 1 | 0
  Sodium, serum-high (hypernatremia) | 0 | 1
  Sodium, serum-low (hyponatremia) | 6 | 1
  Syndromes-Other (Specify) | 1 | 0
  Thrombosis/thrombus/embolism | 2 | 0
  Voice changes/dysarthria | 1 | 0
  Vomiting | 2 | 0
  Weight loss | 1 | 0

ADVERSE EVENTS:
Time Frame: Toxicity assessment was evaluated after each cycle (21 days), up to 2 years.
Description: Only patients with measurable disease at baseline will be included in this analysis.
Groups:
- Ziv-aflibercept + Topotecan: There are total 97 patients in this arm, but only 92 patients with measurable disease at baseline will be included in this analysis.
- Topotecan: There are total 92 patients in this arm, but only 87 patients with measurable disease at baseline will be included in this analysis.
Arm/Group | Ziv-aflibercept + Topotecan | Topotecan
Serious Adverse Events (participants affected / at risk) | 44/92 | 17/87
Other Adverse Events (participants affected / at risk) | 91/92 | 86/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziv-aflibercept + Topotecan (N=92) | Topotecan (N=87)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 3 | 1
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Cardiac General-Other (Cardiac disorders) | 0 | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
SVT and nodal arrhythmia - Atrial flutter (Cardiac disorders) | 1 | 0
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death not associated with CTCAE term - Death NOS (General disorders) | 6 | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 | 0
Pain - Pain NOS (General disorders) | 3 | 0
Syndromes-Other (General disorders) | 1 | 0
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 | 0
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Catheter (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 0 | 1
Infection with unknown ANC - Blood (Infections and infestations) | 0 | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 | 0
AST, SGOT (Investigations) | 1 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 1 | 0
Creatinine (Investigations) | 1 | 0
GGT (gamma-glutamyl transpeptidase) (Investigations) | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 | 0
Platelets (Investigations) | 8 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 8
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Leukoencephalopathy (radiolographic findings) (Nervous system disorders) | 1 | 0
Pain - Head/headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 4 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziv-aflibercept + Topotecan (N=92) | Topotecan (N=87)
Hemoglobin (Blood and lymphatic system disorders) | 64 | 65
Constipation (Gastrointestinal disorders) | 34 | 31
Diarrhea (Gastrointestinal disorders) | 15 | 14
Distention/bloating, abdominal (Gastrointestinal disorders) | 5 | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 7 | 4
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5 | 5
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 34 | 33
Pain - Abdomen NOS (Gastrointestinal disorders) | 13 | 11
Pain - Stomach (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 14 | 17
Edema: limb (General disorders) | 7 | 9
Fatigue (asthenia, lethargy, malaise) (General disorders) | 65 | 56
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 7 | 4
Pain - Chest/thorax NOS (General disorders) | 16 | 12
Pain-Other (General disorders) | 3 | 7
Rigors/chills (General disorders) | 8 | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 12 | 9
AST, SGOT (Investigations) | 14 | 12
Alkaline phosphatase (Investigations) | 17 | 14
Creatinine (Investigations) | 10 | 13
Leukocytes (total WBC) (Investigations) | 52 | 50
Lymphopenia (Investigations) | 16 | 23
Metabolic/Laboratory-Other (Investigations) | 7 | 7
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 53 | 42
Platelets (Investigations) | 70 | 62
Weight loss (Investigations) | 23 | 8
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 22 | 20
Anorexia (Metabolism and nutrition disorders) | 35 | 28
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 6 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 16 | 12
Dehydration (Metabolism and nutrition disorders) | 9 | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 27 | 39
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 19 | 10
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 14 | 21
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 26 | 24
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 14 | 7
Pain - Back (Musculoskeletal and connective tissue disorders) | 17 | 17
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain - Joint (Musculoskeletal and connective tissue disorders) | 5 | 9
Dizziness (Nervous system disorders) | 7 | 16
Neuropathy: sensory (Nervous system disorders) | 8 | 13
Pain - Head/headache (Nervous system disorders) | 18 | 12
Taste alteration (dysgeusia) (Nervous system disorders) | 6 | 5
Confusion (Psychiatric disorders) | 5 | 2
Insomnia (Psychiatric disorders) | 16 | 15
Mood alteration - anxiety (Psychiatric disorders) | 8 | 11
Mood alteration - depression (Psychiatric disorders) | 6 | 6
Proteinuria (Renal and urinary disorders) | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 32
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 38 | 31
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 16 | 4
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 12 | 19
Hypertension (Vascular disorders) | 23 | 2
Hypotension (Vascular disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less